CLINICAL TRIAL: NCT06537414
Title: A Phase 2b, Multi-centre, Randomized, Partially Placebo-controlled, Double-blind Study to Investigate the Safety and Efficacy of Sequential Therapy With Daplusiran/Tomligisiran Followed by Bepirovirsen in Participants With Chronic Hepatitis B Virus on Background Nucleos(t)Ide Analogue Therapy (B-United)
Brief Title: A Study of Sequential Therapy With Daplusiran/Tomligisiran (DAP/TOM) Followed by Bepirovirsen in Participants Living With Chronic Hepatitis B (CHB)
Acronym: B-UNITED
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 218309
Record Dates: First submitted 2024-08-01; First posted 2024-08-05 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B Virus Infection; Hepatitis B
Keywords: Bepirovirsen; B-UNITED; Daplusiran/Tomligisiran; Hepatitis B; Nucleos(t)ide analogue
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment Arm 1A: DAP/TOM + Bepirovirsen (Experimental): Participants with high Hepatitis B surface antigen (HBsAg) level will receive dose level 1 of DAP/TOM in Treatment Stage 1. After DAP/TOM Treatment, eligible participants will receive bepirovirsen in Treatment Stage 2. All participants will continue background NA treatment throughout these treatment stages. After bepirovirsen Treatment Stage, participants will be observed during the NA Only Stage, while maintaining background NA treatment. Eligible participants will then discontinue background NA treatment.
  Interventions: Drug: Daplusiran/Tomligisiran Dose Level 1; Drug: Bepirovirsen
- Treatment Arm 1B: DAP/TOM + Bepirovirsen (Experimental): Participants with high HBsAg level will receive dose level 2 of DAP/TOM in Treatment Stage 1. After DAP/TOM treatment, eligible participants will receive bepirovirsen in Treatment Stage 2. All participants will continue background NA treatment throughout these treatment stages. After bepirovirsen Treatment Stage, participants will be observed during the NA Only Stage, while maintaining background NA treatment. Eligible participants will then discontinue background NA treatment.
  Interventions: Drug: Daplusiran/Tomligisiran Dose Level 2; Drug: Bepirovirsen
- Treatment Arm 2A: DAP/TOM + Bepirovirsen (Experimental): Participants with low HBsAg level will receive dose level 1 of DAP/TOM in Treatment Stage 1. After DAP/TOM treatment, eligible participants will receive bepirovirsen in Treatment Stage 2. All participants will continue background NA treatment throughout these treatment stages. After bepirovirsen Treatment Stage, participants will be observed during the NA Only Stage, while maintaining background NA treatment. Eligible participants will then discontinue background NA treatment.
  Interventions: Drug: Daplusiran/Tomligisiran Dose Level 1; Drug: Bepirovirsen
- Treatment Arm 2B: DAP/TOM + Bepirovirsen (Experimental): Participants with low HBsAg level will receive dose level 2 of DAP/TOM in Treatment Stage 1. After DAP/TOM treatment, eligible participants will receive bepirovirsen in Treatment Stage 2. All participants will continue background NA treatment throughout these treatment stages. After bepirovirsen Treatment Stage, participants will be observed during the NA Only Stage, while maintaining background NA treatment. Eligible participants will then discontinue background NA treatment.
  Interventions: Drug: Daplusiran/Tomligisiran Dose Level 2; Drug: Bepirovirsen
- Treatment Arm 2C: Placebo + Bepirovirsen (Experimental): Participants with low HBsAg level will receive Placebo in Treatment Stage 1. After Placebo treatment, eligible participants will receive bepirovirsen in Treatment Stage 2. All participants will continue background NA treatment throughout these treatment stages. After bepirovirsen Treatment Stage, participants will be observed during the NA Only Stage, while maintaining background NA treatment. Eligible participants will then discontinue background NA treatment.
  Interventions: Drug: Bepirovirsen; Drug: Placebo

INTERVENTIONS:
Drug: Daplusiran/Tomligisiran Dose Level 1 — Daplusiran/Tomligisiran dose level 1 will be administered
  Arms: Treatment Arm 1A: DAP/TOM + Bepirovirsen; Treatment Arm 2A: DAP/TOM + Bepirovirsen
Drug: Daplusiran/Tomligisiran Dose Level 2 — Daplusiran/Tomligisiran dose level 2 will be administered
  Arms: Treatment Arm 1B: DAP/TOM + Bepirovirsen; Treatment Arm 2B: DAP/TOM + Bepirovirsen
Drug: Bepirovirsen — Bepirovirsen will be administered
Drug: Placebo — Placebo will be administered
  Arms: Treatment Arm 2C: Placebo + Bepirovirsen

SUMMARY:
The study is intended to evaluate the efficacy and safety of 2 different doses of DAP/TOM followed by bepirovirsen in participants living with CHB on standard of care nucleos(t)ide analogue (NA) therapy. The study also aims to identify an optimal dose of DAP/TOM for sequenced therapy with bepirovirsen for further clinical development and to assess the contribution of DAP/TOM to the sequential regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 18 years of age at the time of signing the informed consent.
* Documented chronic HBV infection >=6 months prior to Screening AND currently receiving stable NA therapy defined as receiving an NA regimen form at least 6 months prior to Screening and with no planned changes to their stable regimen over the duration of the study.
* Plasma or serum HBsAg concentration >100 international units per milliliter (IU/mL)
* Plasma or serum HBV DNA concentration must be adequately suppressed, defined as plasma or serum HBV DNA <90 IU/mL.
* Alanine aminotransferase <=2* upper limit of normal (ULN)
* Participants who are willing and able to cease their NA treatment in accordance with the protocol.
* Male and Female

Exclusion Criteria:

* Clinically significant abnormalities, aside from chronic HBV infection in medical history (e.g., moderate-severe liver disease other than chronic HBV, acute coronary syndrome within 6 months of screening, major surgery within 3 months of screening, significant/unstable cardiac disease, uncontrolled diabetes, bleeding diathesis coagulopathy) or clinically significant physical examination findings.
* Coinfection with Hepatitis C (cured <12 months at the time of screening), Human immunodeficiency virus or hepatitis D virus.
* History of or suspected liver cirrhosis and/or evidence of cirrhosis.
* Diagnosed or suspected hepatocellular carcinoma.
* History of malignancy within the past 5 years with the exception of specific cancers that are cured by surgical resection (example, skin cancer). Participants under evaluation for possible malignancy are not eligible.
* History of vasculitis or presence of symptoms and signs of potential vasculitis (e.g., vasculitic rash, skin ulceration, repeated blood detected in urine without identified cause), current or history of an autoimmune condition or history/presence of other diseases that may be associated with vasculitis condition (example, systemic lupus erythematosus, rheumatoid arthritis, relapsing polychondritis, mononeuritis multiplex).
* History of extrahepatic disorders possibly related to HBV immune conditions (example, nephrotic syndrome, any type of glomerulonephritis, polyarteritis nodosa, cryoglobulinemia, uncontrolled hypertension).
* History of alcohol or drug abuse/dependence:
* Currently taking, or took within 3 months of screening, any immunosuppressing drugs (example, prednisone), other than a short course of therapy (<=2 weeks) or topical/inhaled steroid use.
* Participants, to whom immunosuppressive treatment (including therapeutic doses of steroids) is contraindicated, should not be considered for enrollment in the study.
* Currently taking, or has taken within 6 months of Screening, any interferon-containing therapy.
* Participants requiring anti-coagulation therapies (example, warfarin, Factor Xa inhibitors) or anti-platelet agents (like clopidogrel or aspirin) unless treatment can safely be discontinued throughout duration of Investigational medicinal product (IMP) treatment, by the discretion of the investigator. Occasional use is permitted.
* Prior hepatitis B treatment with bepirovirsen, DAP/TOM, or another oligonucleotide or small interfering ribonucleic acid (RNA) (siRNA).
* Prior non-hepatitis B treatment with an oligonucleotide or siRNA within 12 months prior to the first dosing day.
* Fridericia's QT correction formula (QTcF) >=450 millisecond (msec) (if single electrocardiogram [ECG] at screening shows QTcF >=450 msec, a mean of triplicate measurements should be used to confirm that participant meets exclusion criterion).
* History of/sensitivity to bepirovirsen, DAP/TOM or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Participants who do not wish to discontinue taking NA therapy for their chronic HBV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving functional cure | Up to 100 Weeks
  The functional cure for Hepatitis B virus (HBV) is defined as sustained suppression (24 weeks or longer) of HBV deoxyribonucleic acid (DNA) <lower limit of quantification (LLOQ) off all HBV treatment and HBsAg not detected with or without Hepatitis B Surface Antibody (HBsAb) after a finite duration of therapy. The number of participants achieving functional cure after discontinuation of all chronic HBV treatments (DAP/TOM, bepirovirsen, and NA treatment) will be reported.

SECONDARY OUTCOMES:
Number of participants achieving functional cure with high Baseline HBsAg level | Up to 100 Weeks
  The functional cure for HBV is defined as sustained suppression (24 weeks or longer) of HBV DNA <LLOQ off all HBV treatment and HBsAg not detected with or without HBsAb after a finite duration of therapy. The number of participants achieving functional cure with high Baseline HBsAg level after discontinuation of all chronic HBV treatments (DAP/TOM, bepirovirsen, and NA treatment) will be reported.
Number of participants achieving functional cure with low Baseline HBsAg level | Up to 100 Weeks
  The functional cure for HBV is defined as sustained suppression (24 weeks or longer) of HBV DNA <LLOQ off all HBV treatment and HBsAg not detected with or without HBsAb after a finite duration of therapy. The number of participants achieving functional cure with low Baseline HBsAg level after discontinuation of all chronic HBV treatments (DAP/TOM, bepirovirsen, and NA treatment) will be reported.
Number of participants achieving functional cure with low Baseline HBsAg level compared against placebo + bepirovirsen arm | Up to 100 Weeks
  The functional cure for HBV is defined as sustained suppression (24 weeks or longer) of HBV DNA <LLOQ off all HBV treatment and HBsAg not detected with or without HBsAb after a finite duration of therapy. The number of participants achieving functional cure with low Baseline HBsAg level after discontinuation of all chronic HBV treatments (DAP/TOM, bepirovirsen, and NA treatment) compared against placebo + bepirovirsen arm will be reported.
Number of participants with undetected HBsAg and HBV DNA <LLOQ | Up to 48 Weeks
  The number of participants with undetected HBsAg and HBV DNA <LLOQ at the end of bepirovirsen treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (69):
- United States (5):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
- Australia (2):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Fitzroy, Victoria
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
- Brazil (4):
  - GSK Investigational Site, Aracaju
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Manaus
  - GSK Investigational Site, São Paulo
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- China (4):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Shanghai
- France (6):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Toulouse
- Germany (3):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Münster
- GSK Investigational Site, Athens, Greece
- Hong Kong (2):
  - GSK Investigational Site, Pokfulam
  - GSK Investigational Site, Shatin
- Italy (7):
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
- Japan (8):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamanashi
- New Zealand (2):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Papatoetoe Auckland
- GSK Investigational Site, Singapore, Singapore
- South Africa (2):
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Reiger Park
- South Korea (4):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, León
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tau-Yuan
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/